CLINICAL TRIAL: NCT00368368
Title: An Open-label Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics/Pharmacodynamics and Safety of GK Activator (2) Following a Single Oral Dose Administration in Patients With Type 2 Diabetes.
Brief Title: A Study of the Effect of Renal Impairment on the Activity of GK Activator (2) in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP19470
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2)
- 2 (Experimental)
  Interventions: Drug: GK Activator (2)
- 3 (Experimental)
  Interventions: Drug: GK Activator (2)

INTERVENTIONS:
Drug: GK Activator (2) — 100mg po

SUMMARY:
This study will investigate the effect of renal impairment on the pharmacokinetics/pharmacodynamics of GK Activator (2) in patients with type 2 diabetes, and will evaluate the effect of renal function on the safety of the drug. Patients will be assigned to treatment groups according to their renal function (normal, moderate renal impairment, or severe renal impairment). After a 1 week washout period from current oral anti-diabetic treatment, all patients will receive a single oral dose of 100mg GK Activator (2), and blood and urine samples will be taken up to 96h post-dose. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes, taken off current sulfonylureas and/or metformin therapy for >=1 week prior to dosing with GK Activator (2);
* normal renal function, or moderate or severe impairment.

Exclusion Criteria:

* type 1 diabetes;
* treatment with insulin or PPAR gamma agonist within 6 months of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Vital signs, adverse events, laboratory parameters. | Throughout study

SECONDARY OUTCOMES:
AUC, Tmax, Cmax, T1/2, CL/F, CLR for GK Activator (2) and metabolite. Glucose Cmax and Cmin, and percentage decrease in glucose from baseline. | Throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (4):
  - Cypress, California
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
- Bratislava, Slovakia